CLINICAL TRIAL: NCT01223651
Title: Performance of Continuous Glucose Monitoring Systems at Altitude.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended awaiting Ministry of Defence ethics approval.
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 10/H0505/73
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Continuous Glucose Monitoring System; Accuracy; Altitude
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGMS at sea level. (Active Comparator): To assess reliability of continuous glucose monitoring system at sea level whilst subject undergo's a hyperinsulinaemic glucose clamp study.
  Interventions: Procedure: two step hyperinsulinaemic glucose clamp study.
- CGMS reliability at simulated 8000 feet. (Active Comparator): To assess reliability of continuous glucose monitoring system at a simulated altitude of 8,000 feet whilst the participant undergo's a hyperinsulinaemic glucose clamp study.
  Interventions: Procedure: two step hyperinsulinaemic glucose clamp study.

INTERVENTIONS:
Procedure: two step hyperinsulinaemic glucose clamp study. — Study participants will have their blood glucose stabilized between 5 - 6 mmol/L by the delivering of a controlled rate insulin/glucose infusion. Participants will have their blood glucose level reduced by conducting a controlled two step hyperinsulinaemic glucose clamp. The clamp procedure will take a total of 120 minutes and will reduce the blood glucose level to below 3 mmol/L. During this time blood tests will be obtained for analysis, physical observations recorded and cognitive function tests performed at regular intervals. Participants will have been fitted at least 12 hours prior to the intervention with 2 real time continuous glucose monitoring systems which will remain in place for the duration of the clamp procedure, however participants will be blinded to their glucose readings.

SUMMARY:
10 healthy volunteers will undergo the controlled lowering of their blood glucose level at sea level and a simulated altitude of 8,000 feet, to test the hypothesis that continuous glucose monitoring system measurement of blood glucose is as accurate at altitude as at sea level.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years.
* No known medical conditions or concomitant medication.

Exclusion Criteria:

* Pregnancy.
* Marine diving in preceding 24 hours.
* Unable to provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of continuous glucose monitoring system (CGMS). | One year.
  To evaluate the accuracy of CGMS for glucose measurement at altitude (8,000 ft) in healthy volunteers.

SECONDARY OUTCOMES:
The effect of altitude on the recognition of hypoglycaemic symptoms. | One year.
  To examine the effect of high altitude (8,000 ft) on the recognition of hypoglycaemia in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Begley, Doctor, Principal Investigator — Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Airforce Base Henlow, Henlow, Bedfordshire
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, Dorset